CLINICAL TRIAL: NCT06320743
Title: Comparison of the Effects of Low and High Flow Sevoflurane Anesthesia on Cerebral and Peripheral Near Infrared Spectroscopy (NIRS) Values in Pediatric Patients
Brief Title: Cerebral and Peripheral Near Infrared Spectroscopy Monitoring in Low and High Flow Anaesthesia in Pediatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Şengül Özmert, Assoc. Prof. MD, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Low Flow Anaesthesia And NIRS
Record Dates: First submitted 2024-03-12; First posted 2024-03-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Child, Only; Inhalation; Vapor; Anesthesia; Cerebral Oxygenation; Cerebral Hypoxia; Peripheral Oxygenation
Keywords: Near Infrared Spectroscopy; Low Flow Sevoflurane Anaesthesia; Pediatric; Cerebral and Peripheral Oxygenation
MeSH Terms: conditions — Respiratory Aspiration; Hypoxia, Brain

STUDY DESIGN:
Intervention Model Description: Cerebral NIRS probe will be attached to the right and left frontotemporal region, and a peripheral NIRS probe will be attached to the inner surface of the forearm and the values will be noted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group LFA (Active Comparator): NIRS probe will be attached to the inner surface of the forearm and cerebral right-left frontotemporal region and the values will be noted. Standard ASA monitoring and induction will be performed. Fresh gas flow will be 4 lt/min, 50% oxygen/air mixture, sevoflurane vaporizer will be turned on at 4%, continue for 10 minutes and then fresh gas flow will be reduced to 0.8 lt/min, sevoflurane the MAK value will be adjusted to be between 0.9-1.1. Alarm limits appropriate to the patient's weight will be determined for all patients, the lower limit of inspired O2 will be set as 30%, the upper limit of inspired CO2 will be set as 5mmHg. If the inspired O2 value drops below 30%, the pulse oximeter peripheral SpO2 drops below 97, and the NIRS values drop by 20%, the oxygen concentration will be increased by 10%. The sevoflurane vaporizer will be turned off 10 minutes before the end of the operation. When the extubation criteria are met, the patient will be extubated.
  Interventions: Device: NIRS ,Ventilation parameters; Device: Oxygen concentration
- Group HFA (Active Comparator): NIRS probe will be attached to the inner surface of the forearm and cerebral right-left frontotemporal region and the values will be noted. Standard ASA monitoring and induction will be performed.Fresh gas flow will be 3lt/min, 50% oxygen/air mixture, and the sevoflurane vaporizer will be turned on at 3%, sevoflurane the MAK value will be adjusted to be between 0.9-1.1. The sevoflurane vaporizer will be turned off the end of the operation. When the extubation criteria are met, the patient will be extubated.
  Interventions: Device: NIRS ,Ventilation parameters

INTERVENTIONS:
Device: NIRS ,Ventilation parameters — NIRS ,Ventilation parameters :
  Until the patient is taken to the operating table and leaves the operating table routine monitoring parameters, BIS values ,cerebral and peripheral NIRS values, until the patient is intubated and extubated ventilation parameters These parameters; 0. min (before induction), 1. min after induction, pre-post intubation, 5. min, 10. min, 20. min, 30. min, 45. min, 60. min, 90. min after connecting to the ventilator. It will then be noted at 1 hour intervals, and finally at the 5th minute after extubation.
Device: Oxygen concentration — Oxygen concentration :
  Alarm limits appropriate to the patient's weight will be determined for all patients, the lower limit of inspired O2 will be set as 30%, the upper limit of inspired CO2 will be set as 5mmHg. If the inspired O2 value drops below 30%, the pulse oximeter peripheral SpO2 drops below 97, and the NIRS values drop by 20%, the oxygen concentration will be increased by 10%
  Arms: Group LFA

SUMMARY:
To investigate the effects of non-invasive cerebral and peripheral NIRS monitoring and low and high flow sevoflurane anaesthesia on cerebral and peripheral NIRS in paediatric patients. To determine the effects of two different flows on these monitoring techniques and thus to facilitate intraoperative patient monitoring and to predict complications (hypoxia) that may occur.

DETAILED DESCRIPTION:
The study will involve American Society of Anesthesiologists Physical Status Classification (ASA) I-III risk group patients, aged between 2 and 12 years, who will under go general anesthesia with a surgical procedure time of 1 hour or more, and who will undergo pediatric surgery, orthopedic and urological surgery, will be included in the study. Preoperative patients' age, gender, height, weight, ASA score and operation type information will be recorded. Patients will be randomized by the sealed envelope method and divided into 2 groups: Low-Flow Anesthesia (LFA) and High-Flow Anesthesia (HFA) groups.

Two groups will undergo NIRS monitoring alongside routine ASA monitoring. Cerebral NIRS probe will be attached to the right and left frontotemporal region, and a peripheral NIRS probe will be attached to the inner surface of the forearm and the basal values will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Between 2-12 years of age, those who are planned to undergo pediatric surgery, orthopedic and urological surgery, and whose procedure time is 1 hour or more
* ASA I-III risk group
* Patients who agreed to be included in the study
* Patients whose informed consent form is approved by their parents will be included in the study.

Exclusion Criteria:

* Patients who do not want to participate in the study
* Patients with ASA score above III
* ASA III patients with decompensated cardiac and pulmonary disease
* Patients with neurological sequelae
* Cases with an operation duration of less than 1 hour
* Patients with contraindications to the use of any anesthetic drugs
* Patients for whom low-flow anesthesia is contraindicated

  * Smoke and gas poisoning
  * Malignant Hyperthermia
  * Septic Shock
  * CO2 absorbent depletion
  * Insufficient oxygen monitoring
* Laparoscopic surgeries
* Patients who develop unexpected intra-operative surgical complications
* Patients whose parents do not approve the informed consent form will not be included in the study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Near infrared spectroscopy (NIRS) | 0., 1., 5., 10., 20., 30., 45., 60., 90.,120.min and every 60 minutes thereafter, finally at the 5th minute after extubation
  Cerebral and peripheral oxygenation will be measured with a NIRS device at low flow and high flow in pediatric patients whose surgical procedure duration is 60 minute or more and who will undergo pediatric surgery, orthopedic and urological surgery under general anesthesia.

SECONDARY OUTCOMES:
Ventilation parameters | 0., 1., 5., 10., 20., 30., 45., 60., 90.,120.min and every 60 minutes thereafter, finally at the 5th minute after extubation
  in the period from intubation to extubation of the patient inspired O2
Ventilation parameters | 0., 1., 5., 10., 20., 30., 45., 60., 90.,120.min and every 60 minutes thereafter, finally at the 5th minute after extubation
  in the period from intubation to extubation of the patient exhaled O2
Ventilation parameters | 0., 1., 5., 10., 20., 30., 45., 60., 90.,120.min and every 60 minutes thereafter, finally at the 5th minute after extubation
  in the period from intubation to extubation of the patient inspire sevoflurane
Ventilation parameters | 0., 1., 5., 10., 20., 30., 45., 60., 90.,120.min and every 60 minutes thereafter, finally at the 5th minute after extubation
  in the period from intubation to extubation of the patient exhaled sevoflurane
Ventilation parameters | 0., 1., 5., 10., 20., 30., 45., 60., 90.,120.min and every 60 minutes thereafter, finally at the 5th minute after extubation
  in the period from intubation to extubation of the patient inspired CO2
Ventilation parameters | 0., 1., 5., 10., 20., 30., 45., 60., 90.,120.min and every 60 minutes thereafter, finally at the 5th minute after extubation
  in the period from intubation to extubation of the patient EtCO2
Ventilation parameters | 0., 1., 5., 10., 20., 30., 45., 60., 90.,120.min and every 60 minutes thereafter, finally at the 5th minute after extubation
  in the period from intubation to extubation of the patient Minimum Alveolar Concentration (MAK)
İntraoperative sevoflurane consumption | Postoperative 5th minute
  Intraoperative sevoflurane consumption in ml will be noted at the end of the case

CONTACTS AND LOCATIONS:
Overall Officials: Sengül Özmert, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No